CLINICAL TRIAL: NCT00806806
Title: A Phase 1 Randomized, Single-blind, Sequential Cohort, Crossover Study to Evaluate the Onset of Action of SKY0402 Following Local Infiltration in Healthy Volunteers
Brief Title: Evaluate the Onset of Action of SKY0402 Following Local Infiltration in Healthy Volunteers
Acronym: TTO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Marius Ardeleanu, MD, Director, Clinical Research, Pacira Pharmaceucticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SKY0402C109
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-08

CONDITIONS: Postoperative Pain Management
Keywords: pain management; postoperative
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SKY0402 (Experimental)
  Interventions: Drug: SKY0402

INTERVENTIONS:
Drug: SKY0402 — Local administration of SKY0402 followed by noxious stimulus
  Arms: SKY0402
Drug: Placebo — Local administration of Placebo followed by noxious stimuli
  Arms: Placebo

SUMMARY:
Given as a single perioperative injection, SKY0402 could provide adequate, continuous, and extended pain relief that could greatly simplify postoperative pain management, reduce the need for repeated administration, and minimize episodes of breakthrough pain.

DETAILED DESCRIPTION:
Subjects will be given either SKY0402 or placebo in response to a noxious stimulus, and the time to onset will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for study entry will meet the following criteria:

* Male or female, ages at least 18 years and not over 55 years.
* Body mass index (BMI) within the range 20.0 to 30.0 kg/m2, inclusive.
* Applies to females only: Female subjects of childbearing potential with a nonsterilized male sexual partner must agree to use a hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device beginning > 30 days prior to the first dosing and continuing until > 7 days after the end of the study. Female subjects who are postmenopausal must have been postmenopausal for > 1 year if they wish not to use contraceptives.
* Good general health, evidenced by a lack of significantly abnormal findings on medical history and screening assessments.
* Pain intensity score of > 30 mm on a VAS after incision and application of an 18% acetic acid solution to nontreated skin (i.e., not infiltrated with any test or control article) at Screening.
* Able and willing to comply with all study visits and procedures, including returning as scheduled for the second treatment visit.
* Able to speak, read, and understand the language of the ICF, study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.
* Willing and capable of providing written informed consent.

Exclusion Criteria:

A subject will not be eligible for the study if he or she meets any of the following criteria:

* A history of hypersensitivity to amide type local anesthetics.
* Pregnancy, nursing, or planning to become pregnant during the course of the study.
* Any current conditions that might interfere with pain assessments, including current pain.
* Conditions of the skin or neurological abnormalities that might alter pain sensitivity. These include excessive scarring, burns, skin grafts, and trauma. Tattoos are permitted.
* A history of keloid formation.
* A coagulopathy or use of medications that might enhance bleeding.
* Use of any of the following medication within the times specified before study drug administration:

  * Long-acting opioid mediations within 3 days.
  * Any opioid medication within 24 hours.
  * Any analgesic medication within 12 hours.
* Consumption of alcohol within 24 hours before either treatment visit.
* Any condition that, in the opinion of the Investigator, renders a subject unsuitable for participation in the study. NOTE: The specific reason(s) for exclusion will be documented in the Screening Log.
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Minor deviations in eligibility criteria are permitted if approved by the Pacira Medical Monitor in agreement with the Investigator prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
time to onset of action | 15 minutes

SECONDARY OUTCOMES:
time to onset | bewteen 15 and 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Marius Ardeleanu, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- The Ohio State University College of Medicine, Dept of Pharmacology, Columbus, Ohio, United States

REFERENCES:
- [Derived] Apseloff G, Onel E, Patou G. Time to onset of analgesia following local infiltration of liposome bupivacaine in healthy volunteers: a randomized, single-blind, sequential cohort, crossover study. Int J Clin Pharmacol Ther. 2013 May;51(5):367-73. doi: 10.5414/CP201775. PMID 23458225